CLINICAL TRIAL: NCT06405932
Title: A Multi-center Randomized Controlled Trial : Study of the Intervention Effect of "a Self-help Mental Fitness Training Camp"on Depression Symptoms During Pregnancy
Brief Title: Study of the Intervention Effect of Self-help Training Camps in Promoting Mental Health Among Perinatal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202451
Record Dates: First submitted 2024-05-05; First posted 2024-05-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mental Health; Perinatal Depression
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Fitness Training Camp (Experimental): The self-help mental fitness training camp, comprising 21 learning modules structured around animated thinking videos, audio, text, and moving images, lasts 21 days. Each learning module is automatically pushed to the intervention group on a daily basis, with an estimated completion time of 30-50 minutes.
  Interventions: Combination Product: Mental Fitness Training Camp
- health education (No Intervention): The control group received routine-care

INTERVENTIONS:
Combination Product: Mental Fitness Training Camp — The Mental Fitness Training camp employs and incorporates core learning content derived from Cognitive Behavioral Therapy and Mindfulness. The program comprises nine thought animations, emotional diary, daily breathing exercises, and pleasure lists.
  Arms: Mental Fitness Training Camp

SUMMARY:
This study was a multi-center randomized controlled trial of an Internet-based self-help mental fitness training camp intervention that included women in early, mid, and late pregnancy with or without psychological distress. A comparison was conducted between the intervention and control groups with regard to depression and anxiety scores during pregnancy and at 42 days postpartum in order to ascertain the efficacy of a self-help mental fitness training camp in preventing negative emotions among perinatal women. In addition, associations between different modes of intervention and maternal and infant outcomes were investigated.

DETAILED DESCRIPTION:
In this study, the principle of "early detection, early diagnosis and early treatment" was used to screen and manage negative emotions such as anxiety and depression in three time windows: early pregnancy, mid-pregnancy and late pregnancy. All weeks from June to December 2024 were randomly divided into intervention and control weeks. Pregnant women were assigned to the intervention or control group according to the week of their visit to the hospital for obstetric examination. The intervention group of pregnant women participated in a three-week program of mental fitness training, while the control group received standard care.

The participants were evaluated on multiple occasions following their enrollment in the study. These evaluations occurred at the baseline stage, immediately following the intervention, during the mid and late stages of pregnancy, and 42 days after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* The gestational week in early pregnancy is 0 to 13 weeks; the gestational week in mid-pregnancy is 14 to 27 weeks; and the gestational week in late pregnancy is 28 to 32 weeks.
* Intention to have children in this pregnancy.
* Ability to understand and complete the questionnaire independently.
* Informed consent and voluntary participation in this study.

Exclusion Criteria:

* Suffering from depression being treated with psychotherapy or medication.
* The presence of a serious mental illness or intellectual disability.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1691 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 0, 3 weeks, 42 days postpartum
  The scale is employed to assess the severity of depression and comprises 10 items, each of which is scored on a 0 to 3 point scale. A total score of 0 to 9 indicates a negative result, 10 to 12 indicates mild depression, 13 to 16 indicates moderate depression, and a score greater than or equal to 17 indicates severe depression.
Generalized Anxiety Disorder | 0, 3 weeks, 42 days postpartum
  The scale is designed to assess the severity of an individual's anxiety symptoms over the past two weeks. It comprises seven entries, each rated on a scale of 0 to 3. A total score of 5 to 9 is indicative of mild anxiety, 10 to 14 of moderate anxiety, and a score of 15 or above of severe anxiety.

SECONDARY OUTCOMES:
Maternal and infant endings | 42 days postpartum
  Maternal pregnancy outcomes and general neonatal outcomes were collected via self-administered scales.
World Health Organization Five-item Well-Being Index | 0, 3 weeks, 42 days postpartum
  The scale in question assesses well-being, with higher total scores representing higher levels of well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Chengli Tang, Study Director — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China